CLINICAL TRIAL: NCT06690762
Title: The Effect of Mobile Technology-Based Education Combined With Relaxation Exercise on Stress, Symptom Severity and Quality of Life in Patients With Irritable Bowel Syndrome.
Brief Title: Relaxation Exercise and Education in Patients With Irritable Bowel Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MAUN-HEM-MC-01
Record Dates: First submitted 2024-11-13; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Irritable Bowel Disease
Keywords: Irritable Bowel Syndrome, Stress, Symptom Severity, Quality of Life, Relaxation
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education (Experimental): It consists of nutrition, physical activity, stress management, relaxation exercises and defecation training.
  Interventions: Other: Education
- Kontrol (No Intervention): no intervention

INTERVENTIONS:
Other: Education — It consists of nutrition, physical activity, stress management, relaxation exercises and defecation training.
  Arms: Education

SUMMARY:
Irritable bowel syndrome (IBS) is a common functional gastrointestinal disorder characterized by chronic recurrent abdominal pain, bloating, changes in bowel habits or bowel movements (1-3). Pharmacological and nonpharmacological methods are used in the treatment of IBS. In addition to lifestyle changes such as dietary changes, physical activity, and stress reduction, relaxation techniques, herbal medicines, and nutritional supplements are important nonpharmacological methods used by IBS patients.

Progressive muscle relaxation exercises (PGE) have been reported to positively affect IBS symptoms, patients' quality of life, anxiety, and depression. PGE training in patients with IBS has been found to improve general health perception, reduce symptom severity, and healthcare costs. (7-9). PGE is a complementary treatment and is among advanced nursing practices (10, 11).

In this study, a mobile application will be developed to educate patients about IBS and PGE. It is thought that this application will reduce the severity of patients' symptoms and increase their quality of life. This study is planned to determine the effects of mobile technology-based training combined with relaxation exercises on stress, symptom severity and quality of life in patients with irritable bowel syndrome.

DETAILED DESCRIPTION:
Definition of Irritable Bowel Syndrome Irritable bowel syndrome is a common functional gastrointestinal disorder characterized by chronic recurrent abdominal pain, bloating, changes in bowel habits or bowel movements. IBS is a chronic, often debilitating, and highly prevalent disorder of the brain-gut interaction that affects 5% to 10% of the population. (8, 12)

Epidemiology of Irritable Bowel Syndrome IBS is a common condition affecting 9% to 23% of the general population, 80% of whom are women, with a significant impact on quality of life and health care costs. Its prevalence is lower in individuals aged 50 years and older. The prevalence of IBS in developed countries has been reported to reach up to 20% of the population.

Population-based epidemiological studies of IBS have shown prevalence rates ranging from 5% to 10% in most countries. It varies between 7% in Southeast Asia and the Middle East studies, 11.8-14.0% in North America, Northern Europe and Australia studies and 15.0-21.0% in Southern Europe, Africa and South America studies. 24 It has been stated that the prevalence of IBS in the general population in China is 6.5%. 25 A national study among middle and high school students in Japan showed that the prevalence of IBS was 18.6%. 26 In a study published in 2020, the prevalence of IBS in the USA, Canada and the United Kingdom was similar between 4.4% and 4.8%.

In our country, studies conducted in İzmir, Sivas, Elazığ and Diyarbakır have stated that the prevalence of IBS varies between 6.2% and 19.1%. The prevalence of IBS in our country varies between 6.3-27% (4-6, 13).

Pathophysiology of Irritable Bowel Syndrome The pathophysiology of IBS is complex, and the pathophysiological mechanisms underlying the syndrome are heterogeneous and not fully understood. However, factors leading to IBS include alterations in brain-gut communication, serotonin metabolism disorders, intestinal motility disorders, visceral hypersensitivity, gastrointestinal infections, altered microbiota, food intolerance, genetics, stress, and psychological factors (8, 13, 14).

Factors such as early life stress, sleep disturbance, maladaptive coping strategies, symptom hypervigilance, and visceral hypersensitivity in IBS patients negatively affect gut-brain communication and increase the likelihood of developing IBS or worsen the severity of IBS (15).

Psychological Factors Psychiatric and psychosomatic conditions often coexist in patients with IBS, and up to 50% of patients meet criteria for a psychiatric diagnosis. A recent meta-analysis of 73 studies concluded that IBS increases an individual's risk of anxiety or depression by three-fold. Several psychosocial factors, including early life experiences, infections, trauma, stress, cultural background, and the level of support an individual receives, are important for IBS (1, 16).

Exacerbation of gastrointestinal symptoms has been found to be more strongly associated with perceived stress in IBS patients than in healthy controls. Stress can activate intestinal mucosal mast cells and stimulate the release of mediators such as serotonin and proinflammatory cytokines, which are responsible for altered bowel sensation and motility. Patients with irritable bowel syndrome often attribute the onset or worsening of visceral pain to stress (8, 17).

Diagnosis of Irritable Bowel Syndrome The pathogenesis of IBS is not clearly understood, and there is no causal biochemical or anatomic disorder that can be used to diagnose IBS. Diagnosis is based on symptoms after exclusion of other GI disorders detected by radiologic or endoscopic testing.

The diagnosis of IBS is symptom-based using the Rome criteria. The Rome IV criteria, derived from a consensus of a multinational group of experts in the field of gut-brain interaction disorders, are used to diagnose IBS for both clinical and research purposes. According to the Rome IV criteria, symptoms must have been present for the past 3 months and have started at least 6 months before diagnosis. Patients with IBS must report symptoms of abdominal pain at least once a week (on average) associated with a change in stool frequency, a change in stool form, and/or a decrease or worsening of abdominal pain associated with defecation (8).

Types of Irritable Bowel Syndrome According to the Rome IV criteria and the predominant stool pattern, IBS patients are divided into four main subtypes: Diarrhea predominant IBS (IBS-D), constipation predominant IBS (IBS-C), IBS with mixed bowel habits (IBS-M), and unclassified IBS. These subgroups are reflected by stool appearance, as assessed by the Bristol Stool Form (BSF) scale, on days with at least one abnormal bowel movement.

Diarrhea predominant IBS (IBS-D); Stools are loose, soft, mushy, or watery in 25% or more of bowel movements, and hard or ball-shaped in less than 25% of bowel movements.

Constipation predominant IBS (IBS-C); Stools are hard or ball-shaped in 25% or more of bowel movements, and watery or loose in less than 25% of bowel movements.

IBS with mixed bowel habits (IBS-M); In 25% or more of the stools, the stool is hard or lumpy and in 25% or more of the stools, the stool is watery like mush.

Unclassified IBS; There is a stool shape that does not fit the other types of IBS (8).

Treatment of Irritable Bowel Syndrome Treatment in IBS includes pharmacological and nonpharmacological treatment methods. Lifestyle interventions such as dietary changes, physical activity and stress reduction represent the most important nonpharmacological approach for patients with IBS.

Considering the influence of psychosocial factors on the clinical symptoms of IBS, practices such as progressive muscle relaxation exercise, meditation, yoga, hypnotherapy, psychoeducation, cognitive-behavioral therapy and acupuncture may be beneficial for patients with IBS (8, 18).

Progressive Relaxation Exercises Progressive muscle relaxation was first described by Jacobson in 1934 as the tensing and releasing of 16 muscle groups. Progressive muscle relaxation exercises involve the voluntary, regular and sequential contraction of 16 muscle groups in the body (hand, forearm, upper arm, forehead, cheek, nose, chin, neck, chest, shoulder, waist, abdomen, stomach, hip, calf, foot, etc.) from head to toe for 5 seconds at maximum along with deep breathing and their relaxation for 10 seconds while focusing on the breath. It is important to explain the relaxation procedures in detail before starting the exercises. This method is repeated for each muscle group and the exercise is completed in an average of 20 minutes. Progressive muscle relaxation exercises reduce muscle tension and provide psychological relief (19, 20). It has been stated that progressive muscle relaxation exercises help patients reduce anxiety and improve their sleep quality because they reduce stress, blood pressure, heart rate, lactic acid production and sensitivity to pain. There are studies examining progressive muscle relaxation exercises in IBS patients in the literature review. A 1993 study found that progressive muscle relaxation exercises caused a 50% reduction in GI symptoms in IBS patients. 14 A randomized controlled trial found that relaxation training reduced IBS symptoms, anxiety, and depression among IBS patients, and improved quality of life. Another study examining the effectiveness of progressive muscle relaxation training in IBS patients found that symptom severity, general health perception, and medical consumption improved significantly immediately after the intervention and also 6 and 12 months after the intervention. In addition, improvements were seen in IBS symptoms, quality of life, and depressive symptoms after progressive muscle relaxation exercises (8, 15, 21, 22).

Nutrition in Irritable Bowel Syndrome Today, it is emphasized that diet and lifestyle recommendations should be the first-step approach in medical nutrition treatment of IBS. Healthy nutrition and lifestyle recommendations are important in IBS management. Many studies report that IBS patients have more irregular eating habits compared to the control group, which can affect motility and contribute to IBS symptoms.

It is recommended that patients with irritable bowel syndrome first change their lifestyle and eating habits. It is important to identify the factors that trigger symptoms and take precautions against them. Dietary changes and eating habits that differ between individuals significantly affect strategies created for improving health and preventing diseases.

A nutrition pyramid specific to IBS was created by Cozma Petrut and his colleagues. The pyramid emphasizes correct eating habits that can improve IBS symptoms and indicates how much of each food group to consume daily. While physical activity and hydration form the basis of the pyramid, fried and processed foods that should be removed from the diet of IBS patients form the top of the pyramid.

Approximately two-thirds of patients with irritable bowel syndrome believe that their symptoms are related to the foods they eat. 50%-70% of these patients report that they cannot tolerate certain foods, 60%-70% report that symptoms worsen after eating, and more than 70% report that foods cause some symptoms. However, despite their widespread use, there is limited data supporting the use of special diets in the treatment of IBS symptoms. It is emphasized that an elimination diet should be focused on in order to determine the role of food intolerance in patients with irritable bowel syndrome. In one study, half of the female IBS patients were found to have improved symptoms after a 3-week diet in which dairy products, citrus fruits, grains, potatoes, coffee, tea, alcohol, and additives were eliminated. Alcohol, caffeine, spicy foods, and fatty foods frequently trigger gastrointestinal symptoms in patients with irritable bowel syndrome. Alcohol affects gastrointestinal motility, absorption, and intestinal permeability; caffeine increases stomach acid secretion and colonic motor activity in healthy individuals. Therefore, regular meal consumption, regular physical activity and good hydration are among the standard recommendations for individuals with IBS. In addition, reducing the intake of spicy foods, alcohol, insoluble fiber, caffeine and fat are among the recommendations. In order to prevent IBS attacks in medical nutrition therapy, approaches such as increasing soluble fiber intake, eliminating foods thought to cause symptoms from the diet and using probiotics/prebiotics are recommended for patients (23).

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older, applied to the polyclinic where the study was conducted,
* Have been diagnosed with IBS according to Rome IV criteria,
* Have a smart phone or computer,
* Have no illness that would prevent them from doing progressive muscle relaxation exercises (heart failure, chronic obstructive pulmonary disease, asthma, pregnant, etc.),

Exclusion Criteria:

* Having communication problems

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-02 (Estimated); Primary Completion 2024-12-06 (Estimated); Study Completion 2025-07-22 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale | three months
  The Perceived Stress Scale (PSS) consists of a total of 14 items. PSS is designed to measure how stressful a person perceives certain situations in their life. Each item is evaluated on a 5-point Likert-type scale ranging from "Never (0)" to "Very often (4)". The 7 items with positive expressions are scored reversely (items 4, 5, 6, 7, 9, 10, and 13). PSS-14 scores range from 0 to 56. A high score indicates a high perception of stress.
IBS symptom severity score | three months
  The IBS symptom severity score (IBS-SSS) was developed to assess the severity of symptoms in IBS. The scale is widely used to monitor the progression and treatment of the disease. The IBS-SSS assesses the severity and duration of abdominal pain (abdominal pain, painful days), abdominal bloating (bloating), satisfaction with bowel habits (bowel habits), and quality of life. The scale consists of a total of 5 questions, each with a score ranging from 0 to 100. The total score of the scale ranges from 0 to 500, with higher scores indicating increased severity of the disease. Scores between 0-74 on the scale are classified as remission, 75-174 as mild, 175-299 as moderate, and 300 and above as severe IBS.
Irritable Bowel Syndrome Quality of Life | three months
  Irritable Bowel Syndrome Quality of Life (IBS QOL) Scale The Irritable Bowel Syndrome Quality of Life (IBS-QOL) Scale was developed to assess the quality of life in patients with Irritable Bowel Syndrome. The 5-point Likert-type scale prepared for IBS patients consists of 34 items and 8 sub-dimensions; The sub-dimensions are mood, activity, body image, health, food avoidance, social response, sexuality and social relationship. The raw scores obtained are evaluated by converting them out of 100 using the formula [Transformed score = (Scale raw score - number of items / maximum possible score - minimum possible score) x 100]. The sub-dimension and total scores of the IBS-QOL scale vary between 0-100. Increasing scale scores indicate that the health-related quality of life of individuals increases.